CLINICAL TRIAL: NCT00622310
Title: Energy Expenditure & Activity During & After Exercise-Induced Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 07-0402; R01DK077088 (NIH)
Record Dates: First submitted 2008-02-21; First posted 2008-02-25 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Exercise (Experimental): Subjects in the EX group will perform supervised exercise 5 d/wk. Exercise will consist primarily of walking on an inclined motor-driven treadmill, but alternate activities will be permitted for 20% of the total exercise sessions (1 of 5 days). Exercise sessions will be preceded by a 5 min warm-up performed at a HR corresponding to 40% of VO2max. The initial exercise duration and intensity at baseline will be 20 minutes at an intensity that elicits a heart rate (HR) corresponding to 60% of VO2max. The target EE will be achieved by a gradual progression of exercise duration and intensity over the first 8 weeks of the exercise program. The target exercise intensity will be the workload corresponding to 75% of VO2max.
  Interventions: Behavioral: Walking exercise
- 2 Walk (Experimental): Subjects in the WALK group will also perform exercise 5 d/wk. Exercise will consist exclusively of walking on level grades, and will be prescribed in two equal duration bouts each day. Subjects in the WALK group will be individually prescribed a walking program based on the EE during moderate intensity walking. The target exercise intensity will be walking speeds corresponding 45% of VO2max.
  Interventions: Behavioral: Walking exercise

INTERVENTIONS:
Behavioral: Walking exercise — Subjects will be randomly assigned to either a structured, vigorous-intensity endurance exercise training program or an intermittent, low-intensity exercise program. Individualized exercise prescriptions will be designed to target an increase of 2500 kcal/wk, and the theoretical weight loss will be approximately 15 pounds (~6.8 kg) during the 6 month intervention.

SUMMARY:
This project is aimed at determining whether an exercise-based weight loss intervention causes a compensation in some component of energy expenditure such that the increase in measured energy expenditure is less than the added exercise. The study will compare two separate exercise interventions to determine if this is influenced by exercise intensity.

DETAILED DESCRIPTION:
The primary aim of this proposed study is to determine how total daily activity thermogenesis (TDAT) and total daily energy expenditure (TDEE) are regulated in obese humans attempting to lose weight and maintain weight loss through exercise. Two exercise interventions will be compared; a structured aerobic exercise program and a walking program. exercise activity thermogenesis (EAT) will be verified, and non-exercise physical activity (NEAT), total daily activity thermogenesis (TDAT), and TDEE will be measured using state-of-the-art technologies. Subjects will be studied during a 6 month intervention period and then during a 6 month follow-up period. It is hypothesized that the walking program will have more favorable effects on TDAT and TDEE during both the intervention and follow-up periods. If the investigators hypotheses are correct, then data from the proposed study could be used to improve the effectiveness of exercise-based weight loss and weight loss maintenance programs.

ELIGIBILITY:
Inclusion Criteria

* Body mass index (BMI) 30-35.0 kg/m2
* Age 18-45 years
* Weight stable (<2 kg weight fluctuation during previous 6 months)
* No regular exercise (> 1 bout of exercise/wk or participation in any sporting activities > 1 hr/wk)
* No self-report of acute or chronic disease (diabetes, heart diseases, and joint problems in particular)
* No current use of prescribed medications
* No plans to relocate within the next year
* No plans for extended travel (> 1 week) within the next 6 months
* No tobacco use

For Females:

* No evidence of amenorrhea (Regular menstrual cycles of 21-35 days)
* Pre-menopausal status (self-report, to be confirmed during screening)
* Pregnancy or lactating within the past year
* No pregnancy or planned pregnancies; sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use one of the following means of contraception: condom, diaphragm, oral or implanted contraceptives, or intrauterine device. Women in exclusive relationships with male partners who have had a successful vasectomy will not be required to use any additional means of birth control.

Exclusion Criteria:

* Claustrphobia;
* Any contraindication(s) to > MRI, e.g. aneurysm, cochlear implant, cardiac pacemaker, or implantable cardiac defibrillator, artificial heart valve, metallic stents, any implantable devices or shunt, weight less than 300 lbs;
* Left Handed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Total daily energy expenditure, assessed using doubly labeled water | Prior to exercise intervention, and 6 months

SECONDARY OUTCOMES:
Total daily activity thermogenesis | Prior to exercise intervention, and 6 months
Body weight and composition | Prior to exercise intervention, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Melanson, PhD, Principal Investigator — University of Colorado Division of Endocrinology, Metabolism, and Diabetes/Division of Geriatrics
Locations (1):
- University of Colorado, School of Medicine, Aurora, Colorado, United States